CLINICAL TRIAL: NCT03785756
Title: A Randomised, Double-Blind, Double-Dummy, Parallel-Group, Multiple-Dose, Active and Placebo-Controlled Efficacy Study of Ibuprofen Prolonged-Release Tablets for the Treatment of Pain After Surgical Removal of Impacted Third Molars
Brief Title: Efficacy of 300 mg Ibuprofen Prolonged-Release Tablets for the Treatment of Pain After Surgical Removal of Impacted Third Molars
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5003601
Record Dates: First submitted 2018-12-17; First posted 2018-12-24 (Actual); Results first posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ibuprofen; Tablets

STUDY DESIGN:
Intervention Model Description: The dental pain model used in this study is a robust and well established postsurgical pain model that produces pain that is predictable in its character, duration, and intensity. The model is widely accepted and has a proven record of assay sensitivity (i.e., separating active drugs from each other, as well as from placebo). The model is frequently used to evaluate NSAID type analgesics. Results from dental pain studies are accepted by the US Food and Drug Administration (FDA) and European authorities and have been widely extrapolated to other general pain conditions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind, double dummy-study. There will be two placebo tablets designed to be comparable to each of the active products (PR and Immediate Release [IR]) in both shape, size, colour and weight. All subject packs have been designed and labelled to ensure blinding is maintained. Subjects, investigators and site staff will all be blind to the treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Prolonged Release Group (Experimental): 2 × 300 mg ibuprofen PR tablets at Hours 0 and 12
  2 × placebo of PR tablets at Hours 8 and 16
  2 × placebo of IR tablets at Hours 0, 8, 12, and 16
  Interventions: Drug: Ibuprofen 300 mg Oral Tablet; Drug: Placebo of PR tablet; Drug: Placebo of IR tablet
- Immediate Release Group (Active Comparator): 2 × 200 mg ibuprofen IR tablets at Hours 0, 8, and 16
  2 × placebo of IR tablets at Hour 12
  2 × placebo of PR tablets at Hours 0, 8, 12, and 16
  Interventions: Drug: Ibuprofen 200 mg Oral Tablet; Drug: Placebo of PR tablet; Drug: Placebo of IR tablet
- Placebo Group (Placebo Comparator): 2 × placebo of PR tablets at Hours 0, 8, 12, and 16
  2 × placebo of IR tablets at Hours 0, 8, 12, and 16
  Interventions: Drug: Placebo of PR tablet; Drug: Placebo of IR tablet

INTERVENTIONS:
Drug: Ibuprofen 300 mg Oral Tablet — 2 × 300 mg tablets at Hours 0 and 12
  Other Names: Prolonged Release Tablet
  Arms: Prolonged Release Group
Drug: Ibuprofen 200 mg Oral Tablet — 2 × 200 mg tablets at Hours 0, 8, and 16
  Other Names: Nurofen, Immediate Release Tablet
  Arms: Immediate Release Group
Drug: Placebo of PR tablet — 2 tablets up to four times in 24 hours
Drug: Placebo of IR tablet — 2 tablets up to four times in 24 hours

SUMMARY:
This is a single centre, randomised, double-blind, double-dummy, parallel group, multiple-dose, active and placebo-controlled efficacy study to evaluate the efficacy and safety of 2×300mg ibuprofen Prolonged Release (PR) tablets in subjects with postoperative dental pain.

DETAILED DESCRIPTION:
This is a single centre, randomised, double-blind, double-dummy, parallel group, multiple-dose, active and placebo controlled efficacy study to evaluate the efficacy and safety of ibuprofen 2 × 300 mg ibuprofen PR tablets in subjects with postoperative dental pain.

Eligible subjects will complete all screening procedures within 28 days before the surgery and randomisation.

At Screening, subjects will provide written informed consent to participate in the study before any protocol specified procedures or assessments are completed. On Day 1, subjects who continue to be eligible for study participation after completing screening procedures and assessments will undergo extraction of 2 or more third molars. At least 1 of the third molars must be a fully or partially bone impacted mandibular molar. If only 2 molars are removed, then they must be ipsilateral.

All subjects will receive local anaesthesia (2% lidocaine with 1:100,000 epinephrine). Nitrous oxide will be allowed at the discretion of the investigator. Subjects who experience moderate to severe pain intensity (a score of ≥5 on a numeric rating scale [NRS] from 0-10 where 0 = no pain, 10 = worst pain ever) within 6 hours after surgery and who continue to meet all study entry criteria will be randomised in a 3:3:1 ratio to receive 2 × 300 mg ibuprofen PR tablets every 12 hours (Q12h), 2 × 200 mg ibuprofen immediate release (IR) tablets every 8 hours (Q8h), or placebo. The randomisation will be stratified by baseline pain category (moderate or severe) using a categorical scale that includes the categories of none (0), mild (1-4), moderate (5-7), and severe (8-10).

Subjects will re-assess their baseline pain intensity using the NRS immediately before receiving study drug (pre-dose, Time 0) and their pain intensity (NRS) and pain relief (5-point categorical scale) at the following time points (pre-dose, if at one of the dosing time points of 0, 8, 12 and/or 16 hours): 15, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, and 24 hours after Time 0; and immediately before each dose of rescue medication, if any. For assessments less than 1 hour apart a window of +/-2 min is allowable whilst for assessments at least 1 hour apart a +/-5 min window is allowable.

The double stopwatch method will be used to record the time to perceptible pain relief and time to meaningful pain relief during the 8 hours following the first dose or until subject takes rescue medication. Subjects will complete a global evaluation of study drug 24 hours (+/- 5 minutes) after Time 0 or immediately before the first dose of rescue medication (whichever occurs first). Vital signs will be recorded after the subject has been in a sitting position for 3 minutes at the following times: before surgery, within 30 minutes before Time 0, 12 and 24 hours after Time 0, and/or immediately before the first dose of rescue medication. Adverse events (AEs) will be monitored and recorded from the time of signing of the informed consent form (ICF) until the Follow-up Visit (or Early Termination Visit). During the 24 hours following Time 0, subjects will complete efficacy and safety assessments. Subjects will remain at the study site overnight and will be discharged on Day 2.

Paracetamol / acetaminophen (1000 mg) will be permitted as the initial rescue medication. Subjects will be encouraged to wait at least 60 minutes after receiving study drug before taking rescue medication. If acetaminophen rescue medication is not effective in relieving the subject's pain, 5 mg oxycodone rescue medication may be administered at the discretion of the investigator.

Subjects are not permitted to take any concomitant medications that might confound assessments of pain relief, such as psychotropic drugs, antidepressants, sedative-hypnotics (other than those permitted for conscious sedation), or other analgesics taken within five times of their elimination half-lives (other than those used at the surgery). Selective serotonin reuptake inhibitors (SSRIs) and serotonin and noradrenaline reuptake inhibitors (SNRIs) are permitted if the subject has been on a stable dose for at least four weeks prior to Visit 1 (screening).

Other restrictions include the following: alcohol use is prohibited from 24 hours before surgery until discharge on Day 2; nothing by mouth from midnight before surgery until 1 hour after surgery; clear liquids only are allowed starting 1 hour after surgery until 1 hour after dosing; 1 hour after dosing, the subject's diet may be advanced according to standard practice.

Upon discharge from the study site, subjects may be prescribed pain medication for use at home according to the standard practice of the study site. On Day 8 (± 2 days), subjects will return to the study site for an abbreviated confirmatory physical assessment and AE assessments.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female ≥ 18 and ≤ 50 years of age.
* Requires extraction of 2 or more third molars. At least 1 of the third molars must be a fully or partially bone impacted mandibular molar. If only 2 molars are removed, then they must be ipsilateral.
* Experiences moderate to severe pain intensity within 6 hours after surgery, as measured by a numeric rating scale (NRS) score of ≥ 5 on a 0-10 scale.
* Has a body weight ≥ 45 kg and a body mass index (BMI) ≤ 35 kg/m².
* Female subjects of child-bearing potential must have been using an acceptable method of contraception for at least 30 days prior to randomisation and be willing to continue use until at least 48 hours post discharge from the clinic.

To be considered not of child-bearing potential, females must be surgically sterile (defined as bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) or post-menopausal (defined as no menses for 12 months without an alternative medical cause).

* Free of clinically significant abnormal findings as determined by medical history, physical examination, vital signs, laboratory tests and ECG.
* Is able to provide written informed consent.
* Is willing and able to comply with study requirements (including diet and smoking restrictions), complete the pain evaluations, remain at the study site overnight, and return for follow up 7 (± 2) days after surgery (Day 8 ± 2 days).

Exclusion Criteria:

* Known hypersensitivity reactions or allergy (e.g., asthma, rhinitis, angioedema or urticaria) in response to nonsteroidal anti-inflammatory drugs (NSAIDs; including ibuprofen), acetylsalicylic acid (aspirin), ingredients of the study drug, or any other drugs used in the study, including anaesthetics and antibiotics that may be required on the day of surgery.
* A history of active or previous peptic ulceration/ haemorrhage, gastrointestinal bleeding or perforation, heart failure, renal or hepatic failure, uncontrolled hypertension, asthma, nasal polyps, or chronic rhinitis.
* Has complications from the tooth extraction or any other clinically significant medical history that, in the opinion of the investigator, would affect the subject's ability to comply or otherwise contraindicate study participation, including but not limited to the following: cardiac, respiratory, gastroenterological, neurological, psychological, immunological, haematological, oncological, or renal disease.
* Has undergone another dental surgery within 60 days prior to the day of surgery.
* A positive urine drugs of abuse screen or alcohol breathalyser test at screening and during the study (with the exception of a positive drugs of abuse screen that is a consequence of permitted prescription medicines).
* If female, has a positive pregnancy test at screening (serum) or on the day of surgery prior to surgery (urine), or is lactating.
* Has known or suspected (in the opinion of the investigator), history of alcoholism or drug abuse within 2 years of screening or evidence of tolerance or physical dependence before dosing with study drug.
* Taking any concomitant medications that might confound assessments of pain relief, such as psychotropic drugs, antidepressants, sedative-hypnotics (other than those permitted for conscious sedation), or other analgesics taken within five times of their elimination half-lives. Selective serotonin reuptake inhibitors (SSRIs) and serotonin and noradrenaline reuptake inhibitors (SNRIs) are permitted if the subject has been on a stable dose for at least four weeks prior to Visit 1 (screening).
* Is considered by the investigator, for any reason (including, but not limited to the risks described as precautions, warnings and contraindications in the current version of the investigator's brochure (IB) for 300 mg ibuprofen PR tablets), to be an unsuitable candidate to receive the study drug.
* Has a history of chronic use (defined as daily use for > 2 weeks) of NSAIDs, opiates, or glucocorticoids (except inhaled nasal steroids and topical corticosteroids), for any condition within 6 months before dosing with study drug.
* Has significant difficulties swallowing capsules or tablets or is unable to tolerate oral medication.
* Subject has received an investigational product or participated in another trial involving a marketed or investigational drug in the 30 days (or for investigational agents with a long half-life, a washout of 5 half-lives) prior to first drug administration (washout period between studies is defined as the period of time elapsed between the last dose of the previous study and first dose for this study), or if the investigator believes that any previous participation in an investigational study would be to the detriment of the safety of the participant or the conduct of the study.
* Enrolment of the Investigator, his / her family members, employees, and other dependent persons.
* Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bertoch, MD, Principal Investigator — JBR Clinical Research
Locations (1):
- JBR Clinical Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Davies NM. Clinical pharmacokinetics of ibuprofen. The first 30 years. Clin Pharmacokinet. 1998 Feb;34(2):101-54. doi: 10.2165/00003088-199834020-00002. PMID 9515184
- [Background] Miles L, Hall J, Jenner B, Addis R, Hutchings S. Predicting rapid analgesic onset of ibuprofen salts compared with ibuprofen acid: Tlag, Tlow, Tmed, and a novel parameter, TCmaxRef. Curr Med Res Opin. 2018 Aug;34(8):1483-1490. doi: 10.1080/03007995.2018.1466697. Epub 2018 Apr 27. PMID 29667449
- [Background] Cooper SA, Desjardins PJ, Turk DC, Dworkin RH, Katz NP, Kehlet H, Ballantyne JC, Burke LB, Carragee E, Cowan P, Croll S, Dionne RA, Farrar JT, Gilron I, Gordon DB, Iyengar S, Jay GW, Kalso EA, Kerns RD, McDermott MP, Raja SN, Rappaport BA, Rauschkolb C, Royal MA, Segerdahl M, Stauffer JW, Todd KH, Vanhove GF, Wallace MS, West C, White RE, Wu C. Research design considerations for single-dose analgesic clinical trials in acute pain: IMMPACT recommendations. Pain. 2016 Feb;157(2):288-301. doi: 10.1097/j.pain.0000000000000375. PMID 26683233
- [Background] Singla NK, Desjardins PJ, Chang PD. A comparison of the clinical and experimental characteristics of four acute surgical pain models: dental extraction, bunionectomy, joint replacement, and soft tissue surgery. Pain. 2014 Mar;155(3):441-456. doi: 10.1016/j.pain.2013.09.002. Epub 2013 Sep 6. PMID 24012952
- See also: Wyeth Consumer Healthcare. (2002). Nonprescription Drug Advisory Committee (NDAC) Meeting on Risks of NSAIDs — https://wayback.archive-it.org/7993/20170405155045/https://www.fda.gov/ohrms/dockets/ac/02/briefing/3882B2_04_Wyeth-Ibuprophen.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Started | 120 | 120 | 40
Completed | 111 | 112 | 35
Not Completed | 9 | 8 | 5

BASELINE CHARACTERISTICS:
Population: One subject in the placebo group withdrew from the study before receiving the allocation intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group | Total
Number analyzed (Participants) | 120 | 120 | 39 | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.6 (2.02) | 19.8 (2.47) | 20.7 (3.13) | 19.8 (2.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 53 | 24 | 149
  Male | 48 | 67 | 15 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 12 | 8 | 37
  Not Hispanic or Latino | 101 | 105 | 30 | 236
  Unknown or Not Reported | 2 | 3 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 3 | 2 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 5 | 2 | 2 | 9
  Black or African American | 2 | 1 | 0 | 3
  White | 107 | 108 | 36 | 251
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 1 | 4 | 0 | 5
Baseline Pain [Mean (Standard Deviation); unit: units on a scale] — Subjects rated their pain using a numeric rating scale (NRS) from 0 (no pain) to 10 (worst pain ever).
  units on a scale | 7.5 (1.23) | 7.6 (1.17) | 7.8 (1.12) | 7.6 (1.19)
Baseline Pain Category [Count of Participants; unit: Participants] — NRS pain scores at baseline (immediately pre-dosing) were categorised as moderate (5-7) and severe (8-10).
  Participants
    Moderate | 63 | 57 | 15 | 135
    Severe | 57 | 63 | 24 | 144
Height [Mean (Standard Deviation); unit: cm] | 168.72 (9.753) | 171.61 (8.517) | 167.85 (6.223) | 169.84 (8.917)
Weight [Mean (Standard Deviation); unit: kg] | 67.99 (13.931) | 73.17 (13.921) | 69.69 (12.041) | 70.46 (13.847)
BMI [Mean (Standard Deviation); unit: kg/m²] | 23.82 (4.085) | 24.79 (4.033) | 24.71 (3.947) | 24.36 (4.057)
Surgery duration [Mean (Standard Deviation); unit: minutes] | 9.2 (4.60) | 9.0 (4.89) | 11.1 (5.81) | 9.4 (4.94)

OUTCOME MEASURES:

1. Primary Outcome: Summed Pain Intensity Difference Over 0 to 12 Hours (SPID12) After Time 0
Description: SPID12 was used to compare the test product (2 × 300 mg ibuprofen PR tablets) and comparator product (2 × 200 mg ibuprofen IR tablets three times a day [TID]) against the placebo product. An 11-point (0-10) numeric rating scale (NRS) for pain was used to assess pain intensity, where a higher score indicates a greater amount of pain. SPID12 was calculated using the summed pain intensity difference (change from Time 0) under the NRS-time curve from 15 minutes through 12 hours calculated using the linear trapezoidal rule and the actual time points, where Time 0 is the time of the first dose of study drug. The minimum value of SPID12 is 0 (no change in pain intensity from Time 0 to 12 hours); the theoretical maximum is 120 (if a patient had a score of 10 [worst pain intensity] at baseline, which decreased to 0 [no pain] at the next time point and remained at 0 after); a higher SPID12 score indicates a better outcome.
Time Frame: 0-12 hours
Population: The ITT Population included all subjects who were treated with study drug and had at least 1 pain assessment after Time 0; it was the primary population for the efficacy analysis.
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale*hours | 51.84 (21.457) | 56.33 (18.769) | 19.11 (24.630)
Statistical Analysis 1: Comparison: Prolonged Release Group vs Placebo Group; The primary efficacy hypothesis was that SPID12 for placebo was equal to SPID12 for ibuprofen 2 × 300 mg PR tablets; Test type: Equivalence — The primary analysis was based on a two-sided test at the significance level of 0.05. The treatment difference is presented with a 95% confidence interval (CI); p < 0.0001, ANCOVA; Estimates from an ANCOVA model with SPID12 score as the dependent variable. Terms for treatment and baseline pain score were included as covariates; Mean Difference (Final Values) = 34.05, 95% CI 2-sided [26.72 to 41.38]

2. Secondary Outcome: Summed Pain Intensity Difference Over 0 to 24 Hours (SPID24) After Time 0
Description: SPID24 was used to compare the test product (2 × 300 mg ibuprofen PR tablets BID) and comparator product (2 × 200 mg ibuprofen IR tablets TID) against the placebo product. An 11-point (0-10) numeric rating scale (NRS) for pain was used to assess pain intensity, where a higher score indicates a greater amount of pain. SPID24 was calculated using the summed pain intensity difference (change from Time 0) under the NRS-time curve from 15 minutes through 24 hours calculated using the linear trapezoidal rule and the actual time points, where Time 0 is the time of the first dose of study drug. The minimum value of SPID24 is 0 (no change in pain intensity from Time 0 to 24 hours); the theoretical maximum is 240 (if a patient had a score of 10 [worst pain intensity] at baseline, which decreased to 0 [no pain] at the next time point and remained at 0 after).
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale*hours | 115.75 (46.146) | 121.90 (37.263) | 64.32 (55.070)

3. Secondary Outcome: Summed Pain Intensity Difference Over 0 to 4 Hours (SPID4) After Time 0
Description: SPID4 was used to compare the test product (2 × 300 mg ibuprofen PR tablets BID) and comparator product (2 × 200 mg ibuprofen IR tablets TID) against the placebo product. An 11-point (0-10) numeric rating scale (NRS) for pain was used to assess pain intensity, where a higher score indicates a greater amount of pain. SPID4 was calculated using the summed pain intensity difference (change from Time 0) under the NRS-time curve from 15 minutes through 4 hours calculated using the linear trapezoidal rule and the actual time points, where Time 0 is the time of the first dose of study drug. The minimum value of SPID4 is 0 (no change in pain intensity from Time 0 to 4 hours); the theoretical maximum is 40 (if a patient had a score of 10 [worst pain intensity] at baseline, which decreased to 0 [no pain] at the next time point and remained at 0 after).
Time Frame: 0-4 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale*hours | 14.68 (9.752) | 16.99 (7.884) | 1.24 (8.346)

4. Secondary Outcome: Summed Pain Intensity Difference Over 0 to 8 Hours (SPID8) After Time 0
Description: SPID8 was used to compare the test product (2 × 300 mg ibuprofen PR tablets BID) and comparator product (2 × 200 mg ibuprofen IR tablets TID) against the placebo product. An 11-point (0-10) numeric rating scale (NRS) for pain was used to assess pain intensity, where a higher score indicates a greater amount of pain. SPID8 was calculated using the summed pain intensity difference (change from Time 0) under the NRS-time curve from 15 minutes through 8 hours calculated using the linear trapezoidal rule and the actual time points, where Time 0 is the time of the first dose of study drug. The minimum value of SPID8 is 0 (no change in pain intensity from Time 0 to 8 hours); the theoretical maximum is 80 (if a patient had a score of 10 [worst pain intensity] at baseline, which decreased to 0 [no pain] at the next time point and remained at 0 after).
Time Frame: 0-8 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale*hours | 33.13 (16.195) | 34.48 (13.001) | 11.00 (14.571)

5. Secondary Outcome: Sum of Total Pain Relief Over 0 to 4 Hours (TOTPAR4) After Time 0
Description: A 5-point categorical Pain Relief Scale (PRS) with choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 was completed in response to the question "How much relief have you had since your starting pain?". Higher scores indicate a better outcome. TOTPAR4 is the total pain relief measured by the PRS from 15 minutes through 4 hours, calculated using the linear trapezoidal rule and the actual time points, where Time 0 is the time of the first dose of study drug. The minimum value of TOTPAR4 is 0 (no pain relief from Time 0 to 4 hours); the theoretical maximum is 16 (if a patient experiences maximum pain relief at all time points after baseline).
Time Frame: 0-4 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale*hours | 8.08 (4.337) | 8.98 (3.365) | 1.98 (3.285)

6. Secondary Outcome: Sum of Total Pain Relief Over 0 to 8 Hours (TOTPAR8) After Time 0
Description: A 5-point categorical Pain Relief Scale (PRS) with choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 was completed in response to the question "How much relief have you had since your starting pain?". Higher scores indicate a better outcome. TOTPAR8 is the total pain relief measured by the PRS from 15 minutes through 8 hours, calculated using the linear trapezoidal rule and the actual time points, where Time 0 is the time of the first dose of study drug. The minimum value of TOTPAR8 is 0 (no pain relief from Time 0 to 8 hours); the theoretical maximum is 32 (if a patient experiences maximum pain relief at all time points after baseline).
Time Frame: 0-8 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale*hours | 18.08 (7.314) | 18.41 (5.764) | 7.89 (5.642)

7. Secondary Outcome: Sum of Total Pain Relief Over 0 to 12 Hours (TOTPAR12) After Time 0
Description: A 5-point categorical Pain Relief Scale (PRS) with choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 was completed in response to the question "How much relief have you had since your starting pain?". Higher scores indicate a better outcome. TOTPAR12 is the total pain relief measured by the PRS from 15 minutes through 12 hours, calculated using the linear trapezoidal rule and the actual time points, where Time 0 is the time of the first dose of study drug. The minimum value of TOTPAR12 is 0 (no pain relief from Time 0 to 12 hours); the theoretical maximum is 48 (if a patient experiences maximum pain relief at all time points after baseline).
Time Frame: 0-12 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale*hours | 28.13 (9.981) | 29.981 (8.538) | 12.76 (9.270)

8. Secondary Outcome: Sum of Total Pain Relief Over 0 to 24 Hours (TOTPAR24) After Time 0
Description: A 5-point categorical Pain Relief Scale (PRS) with choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 was completed in response to the question "How much relief have you had since your starting pain?". Higher scores indicate a better outcome. TOTPAR24 is the total pain relief measured by the PRS from 15 minutes through 24 hours, calculated using the linear trapezoidal rule and the actual time points, where Time 0 is the time of the first dose of study drug. The minimum value of TOTPAR24 is 0 (no pain relief from Time 0 to 24 hours); the theoretical maximum is 96 (if a patient experiences maximum pain relief at all time points after baseline).
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale*hours | 62.32 (20.504) | 64.63 (16.774) | 36.96 (22.153)

9. Secondary Outcome: Summed Pain Relief and Intensity Difference (Sum of TOTPAR and SPID [SPRID]) Over 0 to 4 Hours (SPRID4) After Time 0
Description: The summed pain relief and intensity difference (sum of TOTPAR and SPID [SPRID]) over 0 to 4 hours (SPRID4) was determined by calculating the difference in the PRS at the 4-hour time point and the 0-hour time point (TOTPAR4) and adding this value to the difference in the NRS for pain at the 4-hour time point and the 0-hour time point (SPID4). The minimum value of SPRID4 is 0; the theoretical maximum is 56; a higher SPRID4 score indicates a better outcome.
Time Frame: 0-4 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale*hours | 22.76 (13.870) | 25.97 (11.011) | 3.22 (11.464)

10. Secondary Outcome: Summed Pain Relief and Intensity Difference (Sum of TOTPAR and SPID [SPRID]) Over 0 to 8 Hours (SPRID8) After Time 0
Description: The summed pain relief and intensity difference (sum of TOTPAR and SPID [SPRID]) over 0 to 8 hours (SPRID8) was determined by calculating the difference in the PRS at the 8-hour time point and the 0-hour time point (TOTPAR8) and adding this value to the difference in the NRS for pain at the 8-hour time point and the 0-hour time point (SPID8). The minimum value of SPRID8 is 0; the theoretical maximum is 112; a higher SPRID8 score indicates a better outcome.
Time Frame: 0-8 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale*hours | 51.21 (22.985) | 52.88 (18.156) | 18.89 (19.916)

11. Secondary Outcome: Summed Pain Relief and Intensity Difference (Sum of TOTPAR and SPID [SPRID]) Over 0 to 12 Hours (SPRID12) After Time 0
Description: The summed pain relief and intensity difference (sum of TOTPAR and SPID [SPRID]) over 0 to 12 hours (SPRID12) was determined by calculating the difference in the PRS at the 12-hour time point and the 0-hour time point (TOTPAR12) and adding this value to the difference in the NRS for pain at the 12-hour time point and the 0-hour time point (SPID12). The minimum value of SPRID12 is 0; the theoretical maximum 168; a higher SPRID12 score indicates a better outcome.
Time Frame: 0-12 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale*hours | 79.97 (30.643) | 86.24 (26.260) | 31.87 (33.539)

12. Secondary Outcome: Summed Pain Relief and Intensity Difference (Sum of TOTPAR and SPID [SPRID]) Over 0 to 24 Hours (SPRID24) After Time 0
Description: The summed pain relief and intensity difference (sum of TOTPAR and SPID [SPRID]) over 0 to 24 hours (SPRID24) was determined by calculating the difference in the PRS at the 24-hour time point and the 0-hour time point (TOTPAR24) and adding this value to the difference in the NRS for pain at the 24-hour time point and the 0-hour time point (SPID24). The minimum value of SPRID24 is 0; the theoretical maximum is 336; a higher SPRID24 score indicates a better outcome.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale*hours | 178.07 (64.783) | 186.53 (51.842) | 101.28 (76.562)

13. Secondary Outcome: Number of Subjects With Response to Study Drug
Description: A responder was defined as a subject with ≥30% improvement in pain intensity at the 8-hour assessment without rescue medication during the first 8 hours. An 11-point (0-10) numeric rating scale (NRS) for pain was used to assess pain intensity, where a higher score indicates a greater amount of pain.
Time Frame: 0-8 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
Participants | 81 | 76 | 5

14. Secondary Outcome: Numeric Rating Scale (NRS) Pain Intensity Difference (PID) at Each Time Point After Time 0
Description: An 11-point (0-10) numeric rating scale (NRS) for pain was used to assess pain intensity, where a higher score indicates a greater amount of pain, and the PID (the difference in NRS pain intensity between each time point and Time 0) at each time point was calculated.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale
  PID 15 Minutes Post-dose | 0.4 (0.97) | 0.5 (1.14) | 0.2 (0.99)
  PID 30 Minutes Post-dose | 1.4 (1.79) | 1.5 (1.90) | 0.3 (1.34)
  PID 45 Minutes Post-dose | 2.1 (2.37) | 2.6 (2.25) | 0.3 (1.57)
  PID 1 Hour Post-dose | 2.9 (2.59) | 3.5 (2.51) | 0.4 (2.02)
  PID 1.5 Hours Post-dose | 3.8 (2.76) | 4.4 (2.41) | 0.3 (2.09)
  PID 2 Hours Post-dose | 4.3 (2.78) | 5.0 (2.38) | 0.4 (2.39)
  PID 3 Hours Post-dose | 4.5 (2.81) | 5.2 (2.27) | 0.3 (2.56)
  PID 4 Hours Post-dose | 4.8 (2.92) | 5.2 (2.27) | 0.3 (2.59)
  PID 5 Hours Post-dose | 4.6 (2.79) | 5.0 (2.16) | 0.6 (2.84)
  PID 6 Hours Post-dose | 5.1 (2.10) | 4.8 (2.19) | 3.2 (3.12)
  PID 7 Hours Post-dose | 5.0 (2.25) | 4.3 (2.29) | 3.0 (2.70)
  PID 8 Hours Post-dose | 4.6 (2.32) | 3.6 (2.31) | 3.0 (2.73)
  PID 10 Hours Post-dose | 5.1 (2.10) | 5.4 (2.03) | 2.0 (2.75)
  PID 12 Hours Post-dose | 4.6 (2.21) | 5.6 (1.92) | 2.1 (3.60)
  PID 16 Hours Post-dose | 5.2 (2.34) | 4.8 (2.26) | 3.2 (2.99)
  PID 24 Hours Post-dose | 5.6 (2.20) | 5.9 (1.68) | 3.9 (3.24)

15. Secondary Outcome: Pain Intensity Score at Each Scheduled Time Point After Time 0
Description: Pain intensity score at each scheduled time point will be assessed using a numeric rating scale (NRS) for pain. An 11-point (0-10) numeric rating scale (NRS) for pain was used to assess pain intensity, where a higher score indicates a greater amount of pain.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale
  Pain Intensity Score at Baseline | 7.5 (1.23) | 7.6 (1.17) | 7.8 (1.12)
  Pain Intensity Score 15 Minutes Post-dose | 7.1 (1.59) | 7.1 (1.61) | 7.6 (1.33)
  Pain Intensity Score 30 Minutes Post-dose | 6.1 (2.06) | 6.1 (2.24) | 7.5 (1.62)
  Pain Intensity Score 45 Minutes Post-dose | 5.5 (2.50) | 5.0 (2.57) | 7.6 (1.74)
  Pain Intensity Score 1 Hour Post-dose | 4.7 (2.68) | 4.0 (2.67) | 7.4 (2.06)
  Pain Intensity Score 1.5 Hours Post-dose | 3.8 (2.79) | 3.2 (2.48) | 7.5 (2.08)
  Pain Intensity Score 2 Hours Post-dose | 3.2 (2.79) | 2.6 (2.39) | 7.4 (2.37)
  Pain Intensity Score 3 Hours Post-dose | 2.9 (2.84) | 2.4 (2.26) | 7.6 (2.46)
  Pain Intensity Score 4 Hours Post-dose | 2.7 (2.89) | 2.3 (2.30) | 7.6 (2.52)
  Pain Intensity Score 5 Hours Post-dose | 2.9 (2.88) | 2.6 (2.28) | 7.2 (2.71)
  Pain Intensity Score 6 Hours Post-dose | 2.4 (2.05) | 2.8 (2.16) | 4.7 (2.78)
  Pain Intensity Score 7 Hours Post-dose | 2.5 (2.32) | 3.3 (2.34) | 4.8 (2.53)
  Pain Intensity Score 8 Hours Post-dose | 2.9 (2.46) | 4.0 (2.48) | 4.8 (2.54)
  Pain Intensity Score 10 Hours Post-dose | 2.4 (2.34) | 2.2 (1.92) | 5.8 (2.53)
  Pain Intensity Score 12 Hours Post-dose | 2.9 (2.30) | 2.0 (1.80) | 5.7 (3.18)
  Pain Intensity Score 16 Hours Post-dose | 2.3 (2.26) | 2.8 (2.23) | 4.6 (2.74)
  Pain Intensity Score 24 Hours Post-dose | 1.8 (2.09) | 1.7 (1.53) | 3.9 (3.01)

16. Secondary Outcome: Pain Relief at Each Scheduled Time Point After Time 0
Description: Pain relief score at each scheduled time point after Time 0 was measured using the Pain Relief Scale (PRS). The PRS was used to measure pain relief and is a 5-point categorical scale, with response choices of: none = 0; a little = 1; some = 2; a lot = 3; and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?". Higher scores indicate a better outcome.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
score on a scale
  15 Minutes Post-dose | 0.3 (0.60) | 0.4 (0.67) | 0.3 (0.44)
  30 Minutes Post-dose | 0.9 (0.92) | 1.0 (0.93) | 0.4 (0.72)
  45 Minutes Post-dose | 1.3 (1.10) | 1.6 (1.15) | 0.5 (0.79)
  1 Hour Post-dose | 1.7 (1.22) | 1.9 (1.21) | 0.6 (0.88)
  1.5 Hours Post-dose | 2.1 (1.26) | 2.4 (1.13) | 0.5 (0.88)
  2 Hours Post-dose | 2.3 (1.22) | 2.6 (1.08) | 0.6 (1.00)
  3 Hours Post-dose | 2.5 (1.31) | 2.7 (0.97) | 0.5 (1.00)
  4 Hours Post-dose | 2.6 (1.39) | 2.7 (1.00) | 0.5 (0.97)
  5 Hours Post-dose | 2.5 (1.34) | 2.6 (1.01) | 0.7 (1.10)
  6 Hours Post-dose | 2.7 (0.96) | 2.5 (0.99) | 1.8 (1.29)
  7 Hours Post-dose | 2.7 (1.06) | 2.3 (1.12) | 1.7 (1.21)
  8 Hours Post-dose | 2.5 (1.11) | 2.1 (1.15) | 1.7 (1.23)
  10 Hours Post-dose | 2.7 (1.06) | 2.9 (0.94) | 1.3 (1.16)
  12 Hours Post-dose | 2.5 (1.04) | 2.9 (0.88) | 1.2 (1.27)
  16 Hours Post-dose | 2.8 (1.06) | 2.6 (1.03) | 1.8 (1.34)
  24 Hours Post-dose | 3.0 (0.96) | 3.1 (0.74) | 2.1 (1.43)

17. Secondary Outcome: Peak Pain Relief
Description: Peak pain relief at each time point was measured using the Pain Relief Scale (PRS). The PRS was used to measure pain relief and is a 5-point categorical scale, response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?". Higher scores indicate a better outcome. For each subject, peak pain relief was calculated as the maximum pain relief over all PRS assessments, and summarised by counts (and percentages) for each PRS score. Peak pain relief was calculated from PRS scores that were adjusted for rescue medication usage using windowed worst observation carried forward (WOCF).
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
Participants
  None | 2 | 1 | 0
  A little relief | 2 | 1 | 2
  Some relief | 8 | 3 | 8
  A lot of relief | 49 | 62 | 23
  Complete relief | 59 | 53 | 6

18. Secondary Outcome: Time to Onset of Analgesia (Measured as Time to Perceptible Pain Relief Confirmed by Time to Meaningful Pain Relief) Using Double Stopwatch
Description: Two stopwatches were started immediately after the subject swallowed the study drug. Subjects were instructed to, "Stop the first stopwatch when you first feel any pain relief whatsoever. This does not mean you feel completely better, although you might, but when you first feel any relief in the pain you have now" (perceptible pain relief), and then, "Stop the second stopwatch when you feel the pain relief is meaningful to you" (meaningful pain relief). If the stopwatches were not stopped within 8 hours after Time 0 use of the stopwatches was discontinued. If the subject had meaningful pain relief (i.e., pressed both stopwatches) then time to onset of analgesia was date/time of perceptible pain relief - date/time of the first dose of study drug. Values presented are from Kaplan-Meier estimates.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
Hours | 0.48 [0.42 to 0.53] | 0.47 [0.37 to 0.51] | NA [NA to NA] — Not estimable due to insufficient number of participants with events.

19. Secondary Outcome: Time to First Perceptible Pain Relief
Description: Two stopwatches were started immediately after the subject swallowed the study drug. Subjects were instructed to, "Stop the first stopwatch when you first feel any pain relief whatsoever. This does not mean you feel completely better, although you might, but when you first feel any relief in the pain you have now" (perceptible pain relief). Time to first perceptible pain relief was date/time of the first reported pain relief (any) as assessed by the subject (i.e., when the subject stopped the first stopwatch, irrespective of the second) - date/time of the first dose of study drug. If the stopwatch were not stopped within 8 hours after Time 0, use of the stopwatches was discontinued. Values presented are from Kaplan-Meier estimates.
Time Frame: 0-8 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
Hours | 0.47 [0.09 to 5.11] | 0.46 [0.04 to 3.96] | 1.01 [0.08 to 3.28]

20. Secondary Outcome: Time to Meaningful Pain Relief
Description: Two stopwatches were started immediately after the subject swallowed the study drug. Each subject was instructed, "Stop the second stopwatch when you feel the pain relief is meaningful to you" (meaningful pain relief). Time to meaningful pain relief was the date/time of the first reported meaningful (subjective) pain relief as assessed by the subject (i.e., when the subject stopped the second stopwatch) - date/time of the first dose of study drug. If the stopwatches were not stopped within 8 hours after Time 0 use of the stopwatches was discontinued. Values presented are from Kaplan-Meier estimates.
Time Frame: 0-8 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
Hours | 1.25 [0.21 to 8.00] | 0.99 [0.29 to 8.00] | 2.88 [0.32 to 7.95]

21. Secondary Outcome: Time to Peak Pain Relief
Description: The PRS was used to measure pain relief and is a 5-point categorical scale, with response choices of: none = 0; a little = 1; some = 2; a lot = 3; and complete = 4 to be completed in response to the question "How much relief have you had since your starting pain?". A higher score indicates greater pain. Time to peak pain relief was the time when peak pain relief (PPR) first occurred. Values presented are from Kaplan-Meier estimates.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
Hours | 3.00 [2.03 to 3.97] | 2.02 [1.98 to 3.00] | 5.02 [3.02 to 11.97]

22. Secondary Outcome: Number of Subjects Using Rescue Medication
Description: After randomisation and administration of study drug, paracetamol/acetaminophen (1000 mg) was permitted as the initial rescue medication. Subjects were encouraged to wait at least 60 minutes after receiving study drug before taking rescue medication. If acetaminophen rescue medication was not effective in relieving the subject's pain, 5 mg oxycodone rescue medication was administered at the discretion of the investigator. At the investigator's discretion, repeat doses of rescue medication were also administered as required.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
Participants | 30 | 19 | 32

23. Secondary Outcome: Time to First Use of Rescue Medication (Median and 95% Confidence Interval)
Description: Time to first use of rescue medication, in hours.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
hours | NA [NA to NA] — Median was not reached. | NA [NA to NA] — Median was not reached. | 1.37 [1.20 to 2.38]

24. Secondary Outcome: Time to First Use of Rescue Medication (Hazard Ratios Versus Placebo)
Description: Time to first use of rescue medication, in hours. Values presented are the hazard ratios, calculated from Cox proportional hazards model with treatment group as a categorical factor and baseline pain as a continuous covariate. A hazard ratio of <1 means that when subjects did take rescue medication, subjects in the ibuprofen groups refrained from taking rescue medication for longer than subjects in the placebo group. A hazard ratio of >1 means that when subjects did take rescue medication, subjects in the placebo group refrained from taking rescue medication for longer than subjects in the ibuprofen groups.
Time Frame: 0-24 hours
Population: The ITT Population included all subjects who were treated with study drug and had at least 1 pain assessment after Time 0; it was the primary population for the efficacy analysis.
  The unit of measure is the hazard ratio of the PR and IR Groups versus the Placebo Group; data are not relevant for the Placebo Group.
Measure: Number (95% Confidence Interval); unit: Hazard ratio versus placebo
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
Number analyzed (Participants) | 120 | 120 | 39
Hazard ratio versus placebo | 0.17 [0.10 to 0.29] | 0.10 [0.06 to 0.18] | NA [NA to NA] — Placebo is used as the reference group for the hazard ratio.

25. Other Pre Specified Outcome: Incidence of Treatment Emergent Adverse Events as Assessed by Patient Response to Questions and Spontaneous Reporting of TEAEs
Description: Incidence of treatment emergent adverse events (TEAEs). Data listings will be provided for protocol specified safety data.
Time Frame: 0-10 days
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Vital Signs Measurements - Blood Pressure in mm/Hg
Description: Incidence of changes in vital sign measurements. Descriptive statistics will be provided at each scheduled time point for each treatment group. Changes from Baseline for vital signs will be calculated for each subject.
Time Frame: 0-10 days
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Vital Signs Measurements - Heart Rate in Beats Per Minute
Description: as for outcome 26
Time Frame: 0-10 days
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Vital Signs Measurements - Respiratory Rate in Breaths Per Minute
Description: as for outcome 26
Time Frame: 0-10 days
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Vital Signs Measurements - Body Temperature in ºC
Description: as for outcome 26
Time Frame: 0-10 days
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Global Evaluation of Efficacy Using 5 Point Categorical Scale
Description: Patient's global evaluation of study drug using 5 point categorical scale, response choices of 0 = poor, 1 = fair, 2 = good, 3 = very good, or 4 = excellent to be completed by the patient in response to the question "How effective do you think the study drug is as a treatment for pain?". Subjects will complete the global evaluation of study drug 24 hours after Time 0 or immediately before the first dose of rescue medication (whichever occurs first).
Time Frame: 0-24 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and recorded from the time of signing of the informed consent form until the Follow-up Visit (or Early Termination Visit); a period of up to 30 days. Only treatment-emergent adverse events (those that started or worsened in intensity or relationship to treatment on or after the first dose of study drug) are reported here.
Arm/Group | Prolonged Release Group | Immediate Release Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120 | 0/39
Other Adverse Events (participants affected / at risk) | 11/120 | 15/120 | 12/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolonged Release Group (N=120) | Immediate Release Group (N=120) | Placebo Group (N=39)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 6 (8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (5) | 3 (6)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Puncture site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling face (General disorders) | 0 (0) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Alveolar osteitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (2)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Product administration error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT03785756/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT03785756/SAP_001.pdf